CLINICAL TRIAL: NCT01111643
Title: Longitudinal Strain in Addition to Visual Assessment of Wall Motion for Ruling in Ischemia in the Emergency Room
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: David S. Blondheim, MD, Hillel Yaffe Medical Center
Other Study IDs: 0023-08-HYMC-CTIL
Record Dates: First submitted 2010-04-25; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- I
  Interventions: Device: Echocardiogram

INTERVENTIONS:
Device: Echocardiogram — An echocardiogram will be repeated at every step, from baseline to peak heart rate setting.

SUMMARY:
To assess the utility of technician-based analysis of echocardiograms with longitudinal strain for ruling-in ischemic chest pain in the emergency room, compared to emergency room (ER) physician opinion and expert echocardiographer analysis of wall motion, both the latter blinded to any relevant clinical data .

ELIGIBILITY:
Inclusion Criteria:

* Chest pain
* No indication of acute myocardial infarction

Exclusion Criteria:

* Patients admitted for acute myocardial infarction
* Patients with known coronary artery disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ER because of chest pain with no prior history coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department Hille Yaffe Medical Center, Hadera, Israel